CLINICAL TRIAL: NCT03325439
Title: A Multicenter, Open-Label, Single-Arm Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Brivaracetam in Neonates With Repeated Electroencephalographic Seizures
Brief Title: A Study to Test the Pharmacokinetics, Efficacy, and Safety of Brivaracetam in Newborns With Repeated Electroencephalographic Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated (The study stopped prematurely due to enrolment challenges, the termination was not linked to any safety issues.)
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01349; 2015-002756-27 (EudraCT Number)
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Electroencephalographic Neonatal Seizures
Keywords: Electroencephalographic neonatal seizures; Brivaracetam; Epilepsy; ENS; Newborns; Pharmacokinetic
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brivaracetam (BRV) (Experimental): Exploratory Cohort and Confirmatory Cohorts
  Interventions: Drug: Brivaracetam (BRV) intravenous (iv); Drug: Brivaracetam (BRV) oral

INTERVENTIONS:
Drug: Brivaracetam (BRV) intravenous (iv) — Exploratory Cohort:
  Subjects will be dosed with BRV (0.5 mg/kg twice daily (bid)) according to the sites standard procedures. Treatment with 1 or more of the following antiepileptic drugs (AEDs): phenobarbital (PB), midazolam (MDZ), phenytoin (PHT), levetiracetam (LEV), or lidocaine (LDC) (first-line, second-line, or subsequent treatment) will continue in parallel with BRV treatment.
  Confirmatory Cohort:
  For subjects who enter the Confirmatory Cohorts, for the strength of BRV 1 mg/kg bid (2 mg/kg/day) has been determined based on the Pharmacokinetic (PK) findings of the Exploratory Cohort. Based on further monitoring of PK and safety findings dosing may be adjusted as new data are available. Administration of BRV is proposed as approximately 15-minute intravenous (iv) infusions. Treatment with previous antiepileptic drugs is permitted to continue if the subject is on a stable dose from 1 hour prior to initiation of the BRV treatment.
  Other Names: Briviact
Drug: Brivaracetam (BRV) oral — Subjects can switch from intravenous (iv) to oral brivaracetam (BRV) at any time during the BRV Extension Period
  Other Names: Briviact

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK) of brivaracetam (BRV) in neonates who have seizures that are not adequately controlled with previous antiepileptic drug (AED) treatment, and to identify the optimal BRV dose (Exploratory Cohort) for the treatment of subjects enrolled into the Confirmatory Cohorts of this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation on video-electroencephalography (VEEG) of >= 2 minutes of cumulative electroencephalographic neonatal seizures (ENS), or >=3 identifiable ENS prior to entering the Evaluation Period, despite receiving previous antiepileptic drug treatment for the treatment of electroencephalographic seizures. The occurrence of ENS during an up to 1-hour period must be confirmed either by the local or central VEEG reader prior to drug administration. Preferably, the central VEEG reader should confirm the required ENS
* Subject is male or female and must be at least 34 weeks of corrected gestational age (CGA). In addition, term neonates up to 27 days of postnatal age (PNA) and preterm neonates up to 40 weeks of CGA and 27 days of PNA can be enrolled
* Subject weighs at least 2.3 kg at the time of enrollment
* Subjects with or without concomitant hypothermia treatment

Exclusion Criteria:

Subjects are not permitted to be enrolled in the study if any of the following criteria are met:

* Subject receiving antiepileptic drug (AED) treatment other than phenobarbital, midazolam, phenytoin, levetiracetam (≤60 mg/kg/day), or lidocaine for the treatment of seizures prior to or at the time of enrollment (Confirmatory Cohorts only)
* Subject with seizures responding to any of the following: previous AED treatment immediately prior to BRV treatment, pyridoxine treatment, or correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or hypocalcemia)
* Subject requires extra corporeal membrane oxygenation
* Subject has seizures related to prenatal maternal drug use or drug withdrawal
* Subject has known severe disturbance of hemostasis, as assessed by the Investigator
* Subject has a poor prognosis for survival, as judged by the Investigator
* Subject has 2x upper limit of normal (ULN) of any of the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP), with the following exception:

For subjects with perinatal asphyxia, elevation of AST, ALT or ALP <5x ULN is acceptable, if initial and peak elevation of liver function tests (LFTs) occurs within 5 days after birth, and the time course of LFT elevation is compatible with hepatic injury due to perinatal asphyxia. The determination of ULN will be based on the subject's gestational age (GA) and the site's normal range values for the respective GA

* Subject has direct (conjugated) bilirubin levels >2 mg/dL
* Subject requiring or expected to require phototherapy or exchange transfusion due to elevated bilirubin
* Subject with rapidly increasing bilirubin that may preclude the subject from inclusion in the study at the discretion of the Investigator

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2021-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (12):
- N01349 204, Leuven, Belgium
- N01349 205, Prague, Czechia
- France (2):
  - N01349 207, Lille
  - N01349 206, Paris
- Germany (2):
  - N01349 218, Erlangen
  - N01349 209, Freiburg im Breisgau
- N01349 211, Cork, Ireland
- Italy (3):
  - N01349 212, Messina
  - N01349 213, Parma
  - N01349 256, Roma
- United Kingdom (2):
  - N01349 251, Cambridge
  - N01349 216, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

REFERENCES:
- [Result] Pressler R, Boylan G, Dempsey E, Klotz KA, Krauwinkel W, Will E, Morita D, Floricel F, Elshoff JP, van den Anker J. Pharmacokinetics and safety of brivaracetam in neonates with repeated electroencephalographic seizures: A multicenter, open-label, single-arm study. Epilepsia Open. 2024 Apr;9(2):522-533. doi: 10.1002/epi4.12875. Epub 2024 Jan 11. PMID 38049197
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in May 2019 and concluded in May 2021.
Pre-assignment Details: No eligible study participants were enrolled in the Confirmatory Cohorts. The study stopped prematurely due to enrolment challenges, the termination was not linked to any safety issues. The Participant Flow refers to the All Subjects Screened.
Groups:
- Exploratory Cohort: Participants in this arm received brivaracetam (BRV) 0.5 milligram per kilogram (mg/kg) administered as an intravenous (iv) solution for injection twice daily (bid) during the 48-hour Evaluation Period. An additional 3 doses of BRV (0.5 mg/kg) could have been administered every 12 hours for 48 hours (at the discretion of the Investigator). Treatment with antiepileptic drugs (AEDs) per standard of care (SToC) (first-line, second-line, or subsequent treatment) were continued in parallel with BRV treatment.
Period: Overall Study
Arm/Group | Exploratory Cohort
Started | 9
Treated (Only 6 of 9 participants were treated with BRV.) | 6
Completed | 6
Not Completed | 3
Not completed — Ineligibility | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the All Study Participants Screened Set which consisted of all study participants who had signed the Informed Consent form (ICF) and underwent the study inclusion and exclusion criteria of the current protocol. No eligible study participants were enrolled in the Confirmatory Cohorts. The study stopped prematurely due to enrolment challenges, the termination was not linked to any safety issues.
Arm/Group | Exploratory Cohort
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Corrected gestational age at time of enrollment is reported.
  weeks | 39.2 (1.9)
Age, Customized [Count of Participants; unit: Participants]
  Gestational Age <37 weeks | 2
  Gestational Age >=37 weeks | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8
  Other/mixed | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Brivaracetam (BRV) Following First Dose on Day 1
Description: Pharmacokinetic blood samples were taken 0.5 to 1 hour, 2 to 4 hours, and 8 to 12 hours after the BRV infusion on Day 1 to determine the BRV plasma concentration.
Time Frame: Pharmacokinetic blood samples were taken 0.5 to 1 hour, 2 to 4 hours, and 8 to 12 hours after the BRV infusion on Day 1
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all study participants who provided at least 1 measurable post-Baseline plasma sample (with recorded sampling time) on at least 1 post-Baseline Visit with documented study drug intake times. Each participant was assessed once within the specified time-range and the average of the participants included in the given time-range is presented here. Here, 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Exploratory Cohort
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  0.5-1 hour: number analyzed (Participants) | 5
  0.5-1 hour | 534.2 (15.4)
  2-4 hours | 500.1 (28.2)
  8-12 hours: number analyzed (Participants) | 5
  8-12 hours | 342.7 (13.2)

2. Secondary Outcome: Percentage of Responders to BRV Treatment From Baseline to 3 Hours After the Initial BRV Treatment
Description: A BRV responder was defined as a participant who achieved the following reduction in seizure burden (electroencephalographic neonatal seizures (ENS) in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment:
  At least 80% reduction in nonsevere seizure burden (Nonsevere seizure burden is defined as <=50% seizure activity on video-electroencephalography (VEEG) in all 30-minute timespans), OR At least 50 % reduction in severe seizure burden (Severe seizure burden is defined as >50 % seizure activity on VEEG in any 30-minute timespan). Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to <= 30 minutes, > 30 to <= 60 minutes, >60 to <= 90 minutes, and >90 to <= 120 minutes.
Time Frame: From Baseline to 3 hours after the initial BRV treatment
Population: Efficacy was not evaluated since the study was stopped after the completion of required enrollment of the Exploratory Cohort due to the lack of enrollment of eligible study participants in the Confirmatory Cohorts. Efficacy analyses was planned to be performed on Confirmatory Cohorts only.
Groups:
- Confirmatory Cohort: For the Confirmatory Cohorts, 3 consecutive cohorts were planned to evaluate the efficacy of BRV. However, no study participants were enrolled in the Confirmatory Cohorts due to the lack of enrollment of eligible study participants.
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With at Least 80% Reduction in Nonsevere Seizure Burden From Baseline to 3 Hours After the Initial BRV Treatment
Description: Nonsevere seizure burden was defined as <=50% seizure activity on VEEG in all 30-minute timespans. Seizure burden was measured during the Baseline Period immediately prior to BRV administration and evaluated for a 2-hour period starting 1 hour after the start of initial BRV. Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to <= 30 minutes, > 30 to <= 60 minutes, >60 to <= 90 minutes, and >90 to <= 120 minutes.
Time Frame: From Baseline to 3 hours after the initial BRV treatment
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Severe Seizure Burden From Baseline to 3 Hours After the Initial BRV Treatment
Description: Severe seizure burden was defined as >50% seizure activity on VEEG in any 30-minute timespan. Seizure burden was measured during the Baseline Period immediately prior to BRV administration and evaluated for a 2-hour period starting 1 hour after the start of initial BRV. Timespans of 30 minutes refer to the following intervals within the 2-hour period: 0 to <= 30 minutes, > 30 to <= 60 minutes, >60 to <= 90 minutes, and >90 to <= 120 minutes.
Time Frame: From Baseline to 3 hours after the initial BRV treatment
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Absolute Change in Average Seizure Burden Measured by Continuous Video-electroencephalography (VEEG) From Baseline to the End of the 96-hour Evaluation Period
Description: Seizure burden was measured by continuous video-electroencephalography (VEEG). Baseline seizure burden is defined as seizure burden measured on the continuous VEEG (total electroencephalographic neonatal seizures (ENS) in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.
Time Frame: From Baseline to the end of the 96-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage Change in Average Seizure Burden Measured by Continuous VEEG From Baseline to the End of the 96-hour Evaluation Period
Description: Seizure burden was measured by continuous video-electroencephalography (VEEG). Baseline seizure burden was defined as seizure burden measured on the continuous VEEG (total electroencephalographic neonatal seizures (ENS) in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.
Time Frame: From Baseline to the end of the 96-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of BRV Responders at the End of the 96-hour Evaluation Period
Description: A BRV responder was defined as a participant who achieves the following reduction in seizure burden (electroencephalographic neonatal seizures (ENS) in minutes per hour) without need for rescue medication, compared to the seizure burden measured during the Baseline Period immediately prior to BRV administration, evaluated for a 2-hour period starting 1 hour after the start of initial BRV treatment:
  At least 80% reduction in nonsevere seizure burden (Nonsevere seizure burden is defined as <=50% seizure activity on VEEG in all 30-minute timespans), OR At least 50% reduction in severe seizure burden (Severe seizure burden is defined as >50% seizure activity on VEEG in any 30-minute timespan).
Time Frame: From Baseline to the end of the 96-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Participants Who Are Seizure-free at 24 Hours Following the Start of Initial BRV Treatment, Categorized by Subjects With Nonsevere or Severe Seizure Burden at Baseline
Description: Seizure freedom is defined as 100 % reduction in seizure burden from Baseline.
Time Frame: From Baseline to 24 hours after the initial BRV treatment
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to Reduction in Seizure Burden for BRV Responders
Description: as for outcome 7
Time Frame: From Baseline to the first timepoint when BRV responder criteria are met (up to 96-hour Evaluation Period)
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Seizure Freedom at the End of the Down-Titration Period
Description: Seizure freedom was defined as 100% reduction in seizure burden from Baseline.
Time Frame: From Baseline to the end of the Down-Titration Period (up to 97 days)
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Electroencephalographic Neonatal Seizures (ENS) Frequency Per Hour From Baseline to the End of the 96-hour Evaluation Period
Description: For this study, an ENS was defined as an EEG seizure lasting for at least 10 seconds on VEEG. Baseline seizure burden was defined as seizure burden measured on the continuous VEEG (total ENS in minutes per hour) during a period of up to 1 hour immediately prior to the first administration of study drug.
Time Frame: From Baseline to the end of the 96-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Participants Who Are Seizure-free by Time Interval Over the 96-hour Evaluation Period Following the Start of the Initial BRV Treatment
Description: Seizure freedom was defined as 100% reduction in seizure burden from Baseline.
Time Frame: From 3 hours following the start of the initial BRV treatment to the end of the 96-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

13. Secondary Outcome: Absolute Difference in Clinical Seizures at the End of the 24-hour Evaluation Period From Baseline for Neonates With Motor Seizures at the Time of Inclusion
Description: Seizures was measured by continuous video-electroencephalography (VEEG).
Time Frame: From Baseline to the end of the 24-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

14. Secondary Outcome: Percent Difference in Clinical Seizures at the End of the 24-hour Evaluation Period From Baseline for Neonates With Motor Seizures at the Time of Inclusion
Description: Seizures was measured by continuous video-electroencephalography (VEEG).
Time Frame: From Baseline to the end of the 24-hour Evaluation Period
Population: as for outcome 2
Arm/Group | Confirmatory Cohort
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) as Reported by the Investigator
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment.
Time Frame: Adverse Events were collected from Screening Period until the Safety Follow-Up Visit (up to Day 75)
Population: The All Study Participants Screened Set consisted of all study participants who had signed the ICF and underwent the study inclusion and exclusion criteria of the current protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Exploratory Cohort | Confirmatory Cohort
Number analyzed (Participants) | 9 | 0
percentage of participants | 55.6 |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Screening Period until the Safety Follow-Up Visit (up to Day 75)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered pharmaceutical product that did not necessarily have a causal relationship with this treatment. Safety analysis was done on All Study Participants Screened Set. Only 6 of 9 participants were treated with BRV. No eligible study participants were enrolled in Confirmatory Cohorts. The study stopped prematurely due to enrolment challenges, termination was not linked to any safety issues.
Arm/Group | Exploratory Cohort
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Cohort (N=9)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exploratory Cohort (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Ammonia increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No eligible study participants were enrolled in the Confirmatory Cohorts. The study stopped prematurely due to enrolment challenges, the termination was not linked to any safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03325439/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03325439/SAP_001.pdf